CLINICAL TRIAL: NCT00278876
Title: Phase II Study of Imatinib Mesylate as Adjuvant Treatment in High-relapse Risk Localized Gastrointestinal Stromal Tumors With C-kit Mutation
Brief Title: Adjuvant Imatinib in High-risk Gastrointestinal Stromal Tumor (GIST) With C-kit Mutation
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Asan Medical Center (Other)
Responsible Party: Principal Investigator, Yoon-Koo Kang, Professor, Asan Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AMC0501; CSTI571BKR08
Record Dates: First submitted 2006-01-17; First posted 2006-01-19 (Estimated); Results first posted 2015-07-27 (Estimated); Last update posted 2020-01-07 (Actual); Status verified 2020-01

CONDITIONS: Sarcoma; Gastrointestinal Stromal Tumors
Keywords: GIST; Imatinib; Adjuvant therapy; Kit mutation
MeSH Terms: conditions — Sarcoma; Gastrointestinal Stromal Tumors | interventions — Imatinib Mesylate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- imatinib mesylate (Experimental): patients receiving adjuvant imatinib mesylate
  Interventions: Drug: Imatinib mesylate (Glivec)

INTERVENTIONS:
Drug: Imatinib mesylate (Glivec) — Imatinib mesylate 400mg/day per oral (day 1-28) every 4 weeks

SUMMARY:
The presence of c-kit mutation is an independent poor prognostic factor for relapse in addition to large size (> 5 cm) and high mitotic rate (> 5/50 high power field [HPF]) in localized gastrointestinal stromal tumor (GIST) patients who underwent complete surgical resection. In addition, the localized GIST which had exon 11 c-kit mutation and features of high-risk for relapse according to National Institute of Health (NIH) consensus guideline (tumor size > 10 cm or mitotic count > 10/50 HPF) also have high-risk of relapse. Until recently, there has been no effective therapy for advanced, unresectable GISTs. However, a new agent, imatinib mesylate, has shown promise in the metastatic setting, and c-kit exon 11 mutation is the strongest prognostic factor for better response and survival. It is reasonable to try imatinib in an earlier and minimal residual status especially for patients at higher risk of relapse and a higher probability of response to imatinib.

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven diagnosis of GIST, with positive immunostaining for KIT (CD117)
* Tumor size > 5 cm and mitotic rate > 5/50HPF(High Power Field), or tumor size > 10 cm irrespective of mitotic rate, or mitotic rate > 10/50 HPF irrespective of tumor size.
* Presence of mutation in exon 11 of c-kit gene.
* Surgery performed from 3 weeks to 8 weeks before administration of Imatinib mesylate.
* No evidence of residual macroscopic and microscopic disease after surgery.
* Absence of distant metastases
* No prior radiation therapy, no prior chemotherapy, no prior therapy with Imatinib mesylate, or any other molecular targeted or biological therapy.
* Age 18 yrs or older
* ECOG(Eastern Cooperative Oncology Group electrocorticogram) performance status = 0-2
* No New York Heart Association (NYHA) Class 3~4 cardiac problems
* Absence of severe and/or uncontrolled concurrent medical disease (e.g., uncontrolled diabetes, uncontrolled chronic renal disease, uncontrolled liver disease, including chronic viral hepatitis judged at risk of reactivation, uncontrolled active infection, such as human immunodeficiency virus (HIV) infection, etc.).
* No ongoing pregnancy or nursing..
* No prior, or ongoing other malignancy, except adequately treated basal cell or squamous cell skin cancer, in situ cervical cancer or adequately treated cancer with eradicative intent for which the patient has been continuously disease-free for 5 years.
* No use of coumarin derivatives at the time of treatment start.
* Adequate liver function, as defined by a serum bilirubin < 1.5 x the institutional upper limit of normal (IULN), aspartate aminotransferase (AST) or alanine aminotransferase (ALT) < 2.5 IULN, obtained within 7 days prior to randomization.
* Adequate renal function, as defined by a serum creatinine < 1.5 x IULN, obtained within 7 days prior to randomization.
* Absolute neutrophil count (ANC) > 1.5 x 109/l and a platelet count > 100 x 109/l obtained within 7 days prior to randomization. Baseline hemoglobin > 9 g/dl (this may be achieved by transfusions if needed).
* Absence of any psychological, familial, sociological or geographical condition potentially hampering compliance with the study protocol and follow-up schedule; those conditions should be discussed with the patient before registration in the trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2005-04; Primary Completion 2007-08 (Actual); Study Completion 2011-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yoon-Koo Kang, M.D., Ph.D., Principal Investigator — Asan Medical Center
Locations (4):
- South Korea (4):
  - National Cancer Center, Goyang
  - Asan Medical Center, Seoul
  - Seoul National University Hospital, Seoul
  - Seoul Samsung Medical Center, Seoul

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Forty-eight patients were enrolled at four centers in South Korea between August 2005 and June 2007.
Pre-assignment Details: One patient was excluded from the study before treatment initiation because of metastatic disease.
Groups:
- Imatinib Mesylate: imatinib mesylate 400 mg daily for 2 years
Period: Overall Study
Arm/Group | Imatinib Mesylate
Started | 47
Completed | 38
Not Completed | 9

BASELINE CHARACTERISTICS:
Population: All enrolled patients were included for baseline analysis.
Arm/Group | Imatinib Mesylate
Number analyzed (Participants) | 47
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 35
  >=65 years | 12
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.3 (10.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23
  Male | 24
Region of Enrollment [Number; unit: participants]
  Korea, Republic of | 47

OUTCOME MEASURES:

1. Primary Outcome: 2-year Relapse Free Survival Rate
Time Frame: 2 years
Measure: Number; unit: percentage of participants
Arm/Group | Imatinib Mesylate
Number analyzed (Participants) | 47
percentage of participants | 93.6

2. Secondary Outcome: 2-year Overall Survival Rate
Time Frame: 2 years
Measure: Number; unit: percentage of participants
Arm/Group | Imatinib Mesylate
Number analyzed (Participants) | 47
percentage of participants | 97.9

3. Secondary Outcome: Toxicity Profile
Description: Number of patients who experienced toxicity from study treatment to evaluate the safety and tolerability of adjuvant imatinib
Time Frame: Monitoring of adverse events will be continued for at least 28days following the last dose of study treatment, up to 3 years.
Measure: Number; unit: participants
Arm/Group | Imatinib Mesylate
Number analyzed (Participants) | 47
participants | 47

ADVERSE EVENTS:
Arm/Group | Imatinib Mesylate
Serious Adverse Events (participants affected / at risk) | 0/47
Other Adverse Events (participants affected / at risk) | 47/47
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Imatinib Mesylate (N=47)
Anemia (Blood and lymphatic system disorders) | 40
Leukopenia (Blood and lymphatic system disorders) | 28
Neutropenia (Blood and lymphatic system disorders) | 34
Thrombocytopenia (Blood and lymphatic system disorders) | 17
Edema (Musculoskeletal and connective tissue disorders) | 42
Weight gain (Musculoskeletal and connective tissue disorders) | 10
Dermatitis (Skin and subcutaneous tissue disorders) | 27
Anorexia (Gastrointestinal disorders) | 29
Nausea (Gastrointestinal disorders) | 23
Vomiting (Gastrointestinal disorders) | 17
Constipation (Gastrointestinal disorders) | 5
Diarrhea (Gastrointestinal disorders) | 26
Dyspepsia (Gastrointestinal disorders) | 13
Asthenia (General disorders) | 25
Insomnia (Psychiatric disorders) | 5
Cough (Respiratory, thoracic and mediastinal disorders) | 14
Elevated aspartate aminotransferase (Hepatobiliary disorders) | 12
Elevated alanine transferase (Hepatobiliary disorders) | 13
Hyperbilirubinemia (Hepatobiliary disorders) | 14
Azotemia (Renal and urinary disorders) | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No